CLINICAL TRIAL: NCT03935685
Title: Pilot Study of Mirtazapine for the Dual Treatment of Depression and Temozolomide-Induced Nausea and Vomiting (CINV) in Newly-Diagnosed High-Grade Glioma Patients on Temozolomide Therapy
Brief Title: Pilot Study of Mirtazapine for the Dual Tx of Depression and CINV in High-Grade Glioma Pts on TMZ
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Daniela A. Bota, Associate Dean, Clinical Research, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20194907; UCI 18-83 (Other: CFCCC)
Record Dates: First submitted 2019-04-02; First posted 2019-05-02 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Glioma of Brain
MeSH Terms: interventions — Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- mirtazapine in glioma patients treated with Temozolomide (Experimental): Using the well-known Beck Depression Inventory, we will assess the changes in depression scores from baseline to after four and eight weeks of treatment with mirtazapine. We will also assess the change in nausea, vomiting, and weight at the same time points, and collect information on tolerability of mirtazapine throughout the course of the study.
  Interventions: Drug: Mirtazapine (Remeron)

INTERVENTIONS:
Drug: Mirtazapine (Remeron) — Eligible patients should start Mirtazapine 15mg and stay there unless not tolerated, If there is no improvement in nausea dose can be increased to 30 mg and respectively 45 mg, 4 days apart. If excessive sleep, dose can be doubled. Patients should not take tryptophan while they are part of the study.

SUMMARY:
The purpose of the study is to estimate the ability of mirtazapine to reduce depression, nausea, and vomiting, and maintain weight in depressed glioma patients undergoing Temozolomide (TMZ) therapy. Of equal importance, the investigators will monitor the tolerability of Mirtazapine in these patients over the course of the study.

DETAILED DESCRIPTION:
Research Hypothesis: For glioma patients undergoing TMZ chemotherapy, Mirtazapine will address TMZ-associated nausea and vomiting (CINV) and weight loss in addition to depression. Mirtazapine acts as an antagonist at the 5-HT3 receptor, which may explain its anti-emetic properties. Mirtazapine is also an appetite stimulant, which may help curb the weight loss associated with TMZ chemotherapy.

Specific aim 1: To administer the Beck Depression Inventory to approximately 100 patients meeting the inclusion/exclusion criteria in order to identify at least 36 with clinical depression (defined as total score >= 21).

Specific aim 2: To put at least 36 clinically depressed patients identified in aim one on mirtazapine for eight weeks.

Specific aim 3: To administer the Beck Depression Inventory to patients from aim two at four weeks and at eight weeks of treatment with mirtazapine.

Specific aim 4: To document weight and frequencies of nausea, vomiting, and insomnia among participants over the course of the study.

Specific aim 5: To document adverse events experienced by participants over the course of the study and determine, to the extent possible, if mirtazapine is the cause.

The investigators will:

1. Assess changes in the distribution of depression scores as measured by the Beck Depression Inventory (a self-administered instrument extensively used and validated in glioma studies) from baseline to after eight weeks of treatment with mirtazapine.
2. Assess changes in nausea, vomiting, Sleeping and body weight between baseline and the eight-week follow-up visit,
3. Document the trajectory of changes in depression, nausea, vomiting, and weight over the three study time points (baseline, four-week, and eight-week visit).
4. Lastly, collect information on the tolerability of mirtazapine in our patient population.

Main Research Hypothesis: The investigators hypothesize that the mirtazapine regimen will improve depression scores at eight-weeks, compared to baseline scores. Further, the investigators hypothesize that the mirtazapine regimen will limit the reduction of weight and the incidence of nausea/vomiting and insomnia at eight weeks compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign and date an informed consent document prior to any study related assessments/procedures are conducted.
* Histologically confirmed diagnosis of glioma
* No prior treatment with temozolomide TMZ
* Patient will receive temozolomide TMZ therapy as part of their standard treatment.
* Males and Females ≥18 years of age at the time of signing the informed consent document. Able to understand consent forms and study materials in English
* Willing to use approved methods of contraception for duration of study
* Karnofsy Performance Score (KPS) of at least 60
* Patients should have stopped any anti-depressant medications by standard of care at least a month before enrolling in the trial
* Willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Prior treatment with other chemotherapy drugs for glioma
* Known hypersensitivity to Mirtazapine and 5-HT3 receptor antagonists
* Life expectancy of less than three months
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression level in glioma patients on temozolomide therapy treated with Mirtazapine | 8 weeks
  The assessment is conducted using the Beck Depression Inventory. The scoring scale ranges from 1 to 63. Participants with a baseline depression score of 21 or more will be classified as depressed and will be issued a prescription for mirtazapine. Total depression score between baseline and eight weeks will be compared for each patient. Distributional properties of the data will be assessed using appropriate statistical method to examine whether there is statistically significant improvement or not.
Patient Weight Change | 8 weeks
  To estimate the ability of mirtazapine to maintain weight in depressed glioma patients undergoing Temozolomide (TMZ) therapy. Weight change for each patient between baseline and 8 week will be calculated and analyzed using applicable statistical method.
Frequency and grade of nausea and vomiting in depressed glioma patients on temozolomide therapy treated with Mirtazapine | 8 weeks
  To assess the patient's level of nausea and vomiting on a nausea/vomiting scale of 1 to 7. Lower value indicates less nausea and vomiting; while higher value indicates more nausea and vomiting. Data will be assessed using appropriate statistical method to examine whether there is statistically significant improvement or not.
Incidence of Treatment-Emergent Adverse Events | 8 weeks
  To monitor the adverse event of Mirtazapine over the course of the study. AEs will be graded according to CTCAE V5.

SECONDARY OUTCOMES:
Percentage of adherence to mirtazapine regimen | 8 weeks
  The percentage will be calculated based on patient's pill diary entries. Higher percentage indicates patient is more compliant.
Frequency of dose modifications of mirtazapine | 8 weeks
  The dose of mirtazapine can be adjusted based on patients' conditions and adverse event reports per protocol. This is defined as the number of times that the mirtazapine dose has to be modified for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Bota, MD PHD, Principal Investigator — University of California, Irvine
Locations (1):
- UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No